CLINICAL TRIAL: NCT03155321
Title: The Assessment of Awareness and Implementation of the SAGES Safe Cholecystectomy Program Among Polish Surgeons, as Well as Their Opinion on the Usefulness of the SAGES Safe Cholecystectomy Rules: Increasing the Safety of Cholecystectomy by Popularising the SAGES Safe Cholecystectomy Program
Brief Title: SAGES Safe Cholecystectomy Program in Polish Reality - Awareness, Implementation and Opinion on Usefulness
Status: Terminated | Type: Observational
Why Stopped: Study was complete
Sponsor: Jagiellonian University (Other)
Responsible Party: Principal Investigator, Paweł Bogacki, MD, Jagiellonian University
Other Study IDs: K/ZDS/005504
Record Dates: First submitted 2017-05-12; First posted 2017-05-16 (Actual); Last update posted 2022-04-07 (Actual); Status verified 2022-03

CONDITIONS: Cholelithiasis; Cholecystectomy, Laparoscopic
MeSH Terms: conditions — Cholelithiasis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Polish General Surgeons: The group is formed by active polish general surgeons, both specialists and in training
  Interventions: Other: It's an observational study - no intervention is planned

INTERVENTIONS:
Other: It's an observational study - no intervention is planned — No intervention is planned

SUMMARY:
The study is designed to assess the awareness of the SAGES Safe Cholecystectomy Program among polish surgeons, as well as the degree of implementation of this Program during laparoscopic cholecystectomy performed in Poland. It also gathers the opinion of polish surgeons on usefulness of each of the SAGES Safe Cholecystectomy Rules

DETAILED DESCRIPTION:
The study is based on an anonymous questionnaire that is distributed among polish surgeons across the country. The questionnaire focuses on the demographic data of the surgeon, their experience in years, a few questions regarding their experience in the field of cholecystectomy surgery and questions about whether or not they are familiar with the SAGES Safe Cholecystectomy Program, Teaching Program for the Culture of Safety in Cholecystectomy, as well as Updated Tokyo Guidelines for the management of acute cholangitis and cholecystitis. The questionnaire is available as an appendix. It is then followed by the list of all the Rules of SAGES Safe Cholecystectomy Program with questions about the usefulness of each of the rule, evaluated in form of a 10-point numeric scale (0 - completely useless, 9 - critical).

The collected data will be subject to statistical analysis, the result of which will form the base for creating the Polish Program for Safe Cholecystectomy that will serve to increase the safety of this very common surgical procedure.

ELIGIBILITY:
Inclusion Criteria:

* general surgery specialist or resident registered in Polish National Doctors' Registry
* filled questionnaire on SAGES Safe Cholecystectomy Program

Exclusion Criteria:

* questionnaire not filled properly, missing answers
* declaration of not being either general surgeon specialist of general surgery resident in Poland

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The population is formed by general surgeons in Poland that perform endoscopic cholecystectomy. It is both specialists and residents in training. No age limit was implemented.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Mean usefulness score of each SAGES Safe Cholecystectomy Rule | 01.04.2017 - 31.12.2017
  The usefulness of each rule will be assessed by the participants on a 10-point numeric scale (0 - useless, 9 - critical) which will be part of the questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Jagiellonian University Medical College, Krakow, Małopolska, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bogacki P, Krzak J, Gotfryd-Bugajska K, Szura M. Evaluation of the usefulness of the SAGES Safe Cholecystectomy Program from the viewpoint of the European surgeon. Wideochir Inne Tech Maloinwazyjne. 2020 Mar;15(1):80-86. doi: 10.5114/wiitm.2019.83297. Epub 2019 Mar 4. PMID 32117489